CLINICAL TRIAL: NCT04676191
Title: Single- Center Performance Assessment of a Contactless Sensor for Vital Physiological Parameters Measurement at Rest and Detection of Diagnostic Indices in Sleep Compared to Cardiorespiratory Polygraphy
Brief Title: Validation of a Contactless Vital Signs Measurement Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sleepiz AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: U1111-1248-9457
Record Dates: First submitted 2020-12-09; First posted 2020-12-19 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Sleep Apnea
Keywords: respiration; sleep
MeSH Terms: conditions — Sleep Apnea Syndromes; Respiratory Aspiration | interventions — Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with sleep disorders, cardiorespiratory or neuromuscular disorders (Experimental)
  Interventions: Device: Sleepiz One+; Device: Polysomnography

INTERVENTIONS:
Device: Sleepiz One+ — Simultaneous sleep study with polysomnography and Sleepiz One+
Device: Polysomnography — Simultaneous sleep study with polysomnography and Sleepiz One+

SUMMARY:
The primary aim of this study is to validate the performance of Sleepiz One+ for the measurement of vital physiological parameters in adult population, against a laboratory-based polysomnography. Additionally, the investigators will evaluate Sleepiz One+ ability to identify patients with a high risk of suffering from a sleep-related breathing disorder based on apnea-hypopnea index estimation. Participants will undergo measurement with Sleepiz One+ and a polysomnography device while resting in bed for 20 min as well as during sleep for the duration of the following night.

ELIGIBILITY:
Inclusion Criteria:

* Age >18years
* Ability and consent to undergo electrophysiological routine assessment
* Informed Consent as documented by signature
* Patients diagnosed or suspected to suffer from sleep apnea or any other sleep related disorder or patients suffering from chronic cardiac, respiratory or neuromuscular disorders
* Ambulatory or stationary patients of Klinik Lengg

Exclusion Criteria:

* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Cardiac pacemaker or another implanted electrical device
* Women who are pregnant
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, delirium etc. of the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Respiration rate measurement accuracy agreement | 60 seconds

SECONDARY OUTCOMES:
Binary classification of sleep apnea severity based on the AHI > 15 of Sleepiz One+ compared to results of Domino software and data manually scored by sleep technician | 1 Night
Instantaneous respiration rate agreement between Sleepiz One+ and nasal cannula | 60 seconds
Average respiration rate agreement between Sleepiz One+ and thoracic respiratory effort belt | 1 Night
Average respiration rate agreement between Sleepiz One+ and nasal cannula | 1 Night
Sleep/wake classification agreement between Sleepiz One+ compared to polysomnography (PSG) data manually scored by sleep technician | 60 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz Bujan, Dr. med., Principal Investigator — Klinik Lengg, Zurich
Locations (1):
- Klinik Lengg AG, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No